CLINICAL TRIAL: NCT06635824
Title: A Prospective, Open-Label, Randomized, Phase 3 Trial of Acasunlimab (GEN1046) in Combination With Pembrolizumab Versus Docetaxel in Subjects With PD-L1 Positive Metastatic Non-Small Cell Lung Cancer After Treatment With a PD-1/PD-L1 Inhibitor and Platinum-Containing Chemotherapy (ABBIL1TY NSCLC-06)
Brief Title: Trial to Evaluate Acasunlimab and Pembrolizumab Combination Superiority Over Standard of Care Docetaxel in Non-Small Cell Lung Cancer (ABBIL1TY NSCLC-06)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCT1046-06; 2024-512998-27-00 (EU CTIS Number); jRCT2051240178 (Registry Identifier: Japan Registry of Clinical Trials); 1010602 (Registry Identifier: UK Research Summary Database); NL-OMON57246 (Registry Identifier: NL CCMO)
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: PD-L1-positive, Locally Advanced (Unresectable Stage IIIB/C) or Metastatic NSCLC
Keywords: Lung Cancer; Solid Tumors; PD-L1; 4-1BB
MeSH Terms: conditions — Lung Neoplasms | interventions — pembrolizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Acasunlimab, 100 mg and pembrolizumab, 400 mg will be administered via intravenous (IV) infusion, once every 6 weeks (Q6W) (Cycle length=42 days).
  Interventions: Drug: Acasunlimab; Drug: Pembrolizumab
- Arm B (Active Comparator): Docetaxel, 75 mg/m^2 will be administered via IV infusion, once every 3 weeks (Q3W) (Cycle length=21 days).
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Acasunlimab — IV infusion
  Other Names: GEN1046; DuoBody®-PD-L1×4-1BB
  Arms: Arm A
Drug: Pembrolizumab — IV infusion
  Arms: Arm A
Drug: Docetaxel — IV infusion
  Arms: Arm B

SUMMARY:
This is a multicenter, randomized, open-label, international, Phase 3 trial to evaluate the efficacy and safety of acasunlimab in combination with pembrolizumab versus docetaxel (standard of care) in participants with locally advanced (unresectable stage IIIB/C) or programmed death ligand 1 (PD-L1)-positive metastatic non-small cell lung cancer (NSCLC) who have been treated with programmed cell death protein 1 (PD-1)/PD-L1 inhibitor and platinum-containing chemotherapy, administered either in combination or sequentially in the locally advanced (unresectable stage IIIB/C) or metastatic setting.

DETAILED DESCRIPTION:
The goal of this trial is to determine the efficacy and safety of acasunlimab (an experimental antibody also known as GEN1046 or DuoBody® PDL1x4-1BB) in combination with pembrolizumab (an antibody known as KEYTRUDA®) compared to that of docetaxel (a standard of care chemotherapy). During the trial, the participant's quality of life will also be evaluated using industry-standard scales of measurement. To be eligible, participants must have:

1. non-small cell lung cancer that are locally advanced, unresectable stage IIIB/C or has metastasized (spread)
2. tumors that are positive for the PD-L1 protein (a biomarker that may be predictive of response to therapy)
3. been previously treated with a PD-1/PD-L1-inhibitor and a platinum-containing cancer therapy administered in combination or sequentially (irrespective of the order).

Other eligibility criteria will also apply.

Participants will be assigned to 1 of 2 active therapies, also known as treatment arms, as follows:

* Acasunlimab (100 milligrams [mg]) and pembrolizumab (400 mg) once every 6 weeks (Q6W), or
* Docetaxel 75 milligrams per meter squared (mg/m^2) once every 3 weeks (Q3W).

The estimated trial duration for a participant will vary but may be up to 5 years, consisting of:

* An optional 3-month pre-screening period
* A 28-day screening period
* Up to 2 years of treatment
* A 90-day safety follow-up period
* Post-treatment follow-up.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has histologically or cytologically confirmed locally advanced (unresectable stage IIIB/C) or metastatic NSCLC (stage IV) with known subtype.
* Participant has progressed radiographically on or after receiving:

  * One prior line of therapy (PD-1/PD-L1 inhibitor and platinum-based chemotherapy concomitantly) in the locally advanced (unresectable stage IIIB/C) or metastatic disease setting; OR
  * No more than 2 prior lines of therapy (PD-1/PD-L1 inhibitor and platinum-based chemotherapy sequentially, irrespective of the order) in the locally advanced (unresectable stage IIIB/C) or metastatic disease setting.
* Participant must have positive tumor PD-L1 expression (tumor cells ≥1%) determined prospectively on a tumor sample from the locally advanced (unresectable stage IIIB/C) or metastatic setting at a sponsor-designated central laboratory.
* Participant has measurable disease according to RECIST v1.1 as assessed by the investigator at baseline.
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 within 7 days of Cycle 1 Day 1.
* Participant has a life expectancy of ≥3 months.
* Participant must have adequate organ and bone marrow function, per laboratory test results within 7 days of trial treatment.

Key Exclusion Criteria:

* Documentation of known targetable epidermal growth factor receptor (EGFR) sensitizing mutations, anaplastic lymphoma kinase (ALK), RET proto-oncogene (RET), ROS proto-oncogene 1; receptor tyrosine kinase (ROS1) rearrangement, Kirsten rat sarcoma virus (KRAS), B-Raf proto-oncogene (BRAF) mutations, and MET proto-oncogene; receptor tyrosine kinase (MET) exon 14 skipping mutations/MET amplification. NOTE: MET amplification testing is optional based on local availability of the test.

  * Participants with known KRAS/BRAF mutations are eligible for the trial if they do not have access to targeted therapies.
* Participants with newly identified, untreated or unstable or symptomatic central nervous system (CNS) metastases or history of carcinomatous meningitis.
* Prior treatment with docetaxel for NSCLC.
* Prior treatment with a 4-1BB (CD137) targeted agent, any type of antitumor vaccine, autologous cell immunotherapy, or any unapproved immunotherapy.
* Treatment with an anticancer agent within 28 days prior to the first dose of trial treatment.

Note: Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 5 years
  OS is defined as the time from date of randomization to date of death due to any cause.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 5 years
  PFS is defined as the time from the date of randomization to the date of the first documented progression or death due to any cause, whichever occurs first based on response evaluation criteria in solid tumors (RECIST) version 1.1 as assessed by the investigator.
Confirmed Overall Response Rate (ORR) | Up to approximately 5 years
  Confirmed ORR is defined as the proportion of participants with best overall response (BOR) of complete response (CR) or partial response (PR) based on RECIST v1.1 as assessed by the investigator.
Duration of Response (DOR) | Up to approximately 5 years
  DOR is defined as the time from the onset date of response to the date of the first documented progression or death due to any cause based on RECIST v1.1 as assessed by the investigator.
Number of Participants With Adverse Events (AEs) | From first dose until the end of the study (approximately 5 years)
Time to Treatment Discontinuation Due to AE | From first dose until the end of the study (approximately 5 years)
Plasma Concentration of Acasunlimab | Predose and postdose at multiple timepoints in Cycles 1-4, then every other cycle starting Cycle 5 (Cycle length=42 days), up to approximately 5 years
Number of Participants With Anti-drug Antibodies (ADAs) to Acasunlimab | Up to approximately 5 years
  Serum samples will be analyzed using validated, specific, and sensitive immunoassay method. Samples will be screened for ADAs binding to acasunlimab and the titer of confirmed positive/negative samples will be reported.
Change From Baseline in Functional Assessment of Cancer Therapy Item GP5 (FACIT-GP5; Version 4) Score | Baseline up to approximately 2 years
  Participant's global assessment of treatment tolerability will be assessed by FACIT-GP5. FACIT-GP5 asks participants to rate their agreement with the following statement, "I am bothered by side effects of treatment" in the past 7 days. Responses will be captured on a 5-point Likert scale ranging from 0 to 4 indicating 0 as not at all to 4 as very much bothered by side effects.
Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to approximately 2 years
  The PRO-CTCAE allows participants to report on the frequency, severity, and interference of patient-reported symptoms. For each AE, there are between one and three items to assess the frequency, severity, and/or interference with activities related to that AE. All PRO-CTCAE responses will be scored from 0 to 4 for frequency indicating (0= never to 4= almost constantly), severity (0= none to 4= very severe) and interference with usual or daily activities (0= not at all to 4= very much).

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (245):
- United States (36):
  - Arizona Blood and Cancer Specialists, Tucson, Arizona
  - Usc Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente Vallejo Medical Center, Vallejo, California
  - Ocala Oncology Center P.L., Ocala, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Piedmont Cancer Institute Atlanta, Atlanta, Georgia
  - Piedmont Cancer Institute - Sandy Springs (Atlanta) Office, Atlanta, Georgia
  - Piedmont Cancer Institute - Fayetteville Office, Fayetteville, Georgia
  - Piedmont Cancer Institute - Newnan Office, Newnan, Georgia
  - Piedmont Cancer Institute - Stockbridge Office, Stockbridge, Georgia
  - Kaiser Foundation Hospitals, Honolulu, Hawaii
  - University of Illinois, Chicago, Illinois
  - Community Cancer Center East Medical Oncology Hematology, Indianapolis, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Pikeville Medical Center, Pikeville, Kentucky
  - Washington University School of Medicine, St Louis, Missouri
  - St. Francis Hospital - Grand Island, Grand Island, Nebraska
  - Oncology Hematology West, Omaha, Nebraska
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Stony Brook University Medical Center|University Medical Center, Stony Brook, New York
  - Novant Health Pharmacy, Charlotte, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Parkridge Medical Center, Chattanooga, Tennessee
  - University of Tennessee Medical Center Cancer Institute, Knoxville, Tennessee
  - Midtown Tennessee Oncology, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology-Austin Central, Austin, Texas
  - South Austin Cancer Ctr, Austin, Texas
  - University of Virginia Hematology and Oncology, Charlottesville, Virginia
  - Cancer Institute At Swedish Med Ctr, Seattle, Washington
- Argentina (6):
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Centro de Investigacion Pergamino S.A., Pergamino, Buenos Aires
  - Instituto Medico Especializado Alexander Fleming, Buenos Aires, Ciudad Autonoma Buenos Aires
  - Sanatorio Parque S.A., Rosario, Santa Fe Province
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Investigaciones CORI S.R.L., La Rioja
- Australia (8):
  - Chris OBrien LifeHouse, Camperdown, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Gold Coast Hospital, Southport, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Sir Charles Gairdner Hospital, Perth, Western Australia
  - St John of God Subiaco Hospital, Subiaco, Western Australia
  - St Vincent's Hospital Melbourne, Fitzroy
  - Ballarat Oncology & Haematology Service, Wendouree
- Austria (4):
  - Kepler Universitatsklinikum Med Campus III, Linz
  - LKH - Rankweil, Rankweil
  - Standort Penzing der Klinik Ottakring, Vienna
  - Wiener Gesundheitsverbund - Klinik Floridsdorf, Vienna
- Belgium (8):
  - C. H. U. St-Pierre, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Bruxelles, Brussels
  - Grand Hôpital de Charleroi, Gilly
  - Jessa Ziekenhuis Hospital, Hasselt
  - CHU de Liège, Liège
  - AZ Sint-Maarten, Mechelen
  - AZ Delta, Roeselare
- Brazil (14):
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - MultiHemo Servicos Medicos, Recife, Pernambuco
  - Instituto D'Or Pesquisa e Ensino - Rio de Janeiro, Rio de Janeiro, Rio Do Janeiro
  - Hospital de Clinicas de Ijui, Ijuí, Rio Grande do Sul
  - Centro Gaucho Integrado - Mae de Deus Center, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande Do Su
  - Clínica de Neoplasias Litoral Ltda., Itajaí, Santa Catarina
  - BP A Beneficencia Portuguesa de Sao Paulo, São Paulo, São Paulo
  - Centro Paulista de Oncologia S.A., São Paulo, São Paulo
  - Hospital Sirio-Libanes, São Paulo, São Paulo
  - Oncoclínicas do Brasil Serviços Médicos SA, Belo Horizonte
  - Hospital Ernesto Dornelles, Porto Alegre
  - Oncoclínicas Rio de Janeiro, Rio de Janeiro
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André
- Bulgaria (6):
  - MHAT Heart and Brain - Pleven, Pleven
  - Complex Oncology Center - Plovdiv, EOOD, Plovdiv
  - MHAT "Serdika", EOOD, Sofia
  - MHAT for women's health - Nadezhda, OOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - UMHAT 'SofiaMed', OOD, Sofia
- Canada (3):
  - William Osler Health System-Brampton Civic Hospital|William Osler Health System, Brampton, Ontario
  - Princess Margaret Cancer Centre - University Health Network, Toronto, Ontario
  - MUHC - Jewish General Hospital, Montreal, Quebec
- Chile (4):
  - FALP - Fundación Arturo López Pérez, Providencia
  - Centro de Investigacion Clinica Bradford Hill, Santiago
  - IRAM - Instituto de Radio Medicina, Santiago
  - Oncocentro APYS, Viña del Mar
- Croatia (4):
  - General Hospital Dubrovnik, Dubrovnik
  - Specialty Hospital Medico, Rijeka
  - Department for Pulmonary Diseases University Hospital Centre Zagreb, Zagreb
  - Sestre milosrdnice University Hospital Center, Zagreb
- Estonia (2):
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- France (19):
  - Institut Paoli Calmettes, Marseille, Bouches-du-Rhône
  - Institut Bergonié, Bordeaux, Gironde
  - Clinique Belharra, Bayonne, Pyrenees Atlantiques
  - Institut Sainte Catherine, Avignon, Vaculuse
  - Institut Gustave Roussy, Villejuif, Val De Marne
  - CHU Angers - Hôpital Larrey, Angers
  - Centre Hospitalier de la côte Basque, Bayonne
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Centre Hospitalier Intercommunal de Creteil (CHIC), Créteil
  - Hopital Albert Calmette - CHU Lille, Lille
  - Centre Léon Bérard, Lyon
  - Assistance Publique-Hôpitaux de Marseille, Marseille
  - CH de Mulhouse - Hôpital Emile Muller, Mulhouse
  - Hôpital Privé du Confluent, Nantes
  - Hopital Saint Joseph - Paris, Paris
  - Institut Curie, Paris
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - ICO - Site René Gauducheau, Saint-Herblain
  - Hôpital Sainte Musse, Toulon
- Germany (13):
  - Klinikum Esslingen GmbH, Esslingen am Neckar, Baden-Wurttemberg
  - Thoraxklinik Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg
  - Universitaetsmedizin Goettingen, Göttingen, Lower Saxony
  - MHH Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Johannes Gutenberg University Mainz, Mainz, Rhineland-Palatinate
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - MVZ Martha-Maria Halle-Doelau, Halle, Saxony-Anhalt
  - LungenClinic Grosshansdorf GmbH, Großhansdorf, Schleswig-Holstein
  - Evangelische Lungenklinik Berlin, Berlin
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Vivantes Klinikum Neukoelln, Berlin
  - Vivantes Klinikum Spandau, Berlin
  - Asklepios Klinik Harburg, Hamburg
- Greece (7):
  - Alexandra General Hospital, Athens
  - Henry Dunant Hospital Center, Athens
  - University General Hospital Attikon, Athens
  - University General Hospital of Heraklion, Heraklion
  - University General Hospital of Larissa, Larissa
  - Bioclinic Thessaloniki, Thessaloniki
  - Interbalkan Hospital of Thessaloniki, Thessaloniki
- Hungary (2):
  - Orszagos Koranyi Pulmonologiai Intezet, Budapest
  - Bács-Kiskun County Hospital BKMK, Kecskemét
- Ireland (6):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - St James's Hospital, Dublin
  - St Vincent's University Hospital, Dublin
  - University Hospital Limerick, Limerick
  - Waterford Regional Hospital, Waterford
- Italy (14):
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Milano
  - Istituto Clinico Humanitas, Rozzano, Milano
  - AOU Università degli Studi della Campania "Luigi Vanvitelli", Naples, Napoli
  - IRCCS Centro di Riferimento Oncologico, Aviano, Pordenone
  - IRCCS Policlinico Universitario Agostino Gemelli, Rome, Roma
  - AOU San Luigi Gonzaga, Orbassano, Torino
  - ASST Papa Giovanni XXIII, Bergamo
  - Istituto di Candiolo, Candiolo
  - Istituto Nazionale per la Ricerca sul Cancro di Genova, Genova
  - IRCCS Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori IRST, Meldola
  - IRCCS Istituto Nazionale dei Tumori, Milan
  - Ospedale Santa Maria delle Croci, Ravenna
  - Regina Elena National Cancer Institute, Roma
  - CRC - Centro Ricerche Cliniche di Verona S.r.l., Verona
- Japan (22):
  - Shikoku Cancer Center, Matsuyama, Ehime
  - JCHO Kyushu Hospital, Kitakyushu-shi, Fukuoka
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Kobe Minimally Invasive Cancer Center, Kobe, Hyōgo
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Juntendo University Hospital, Bunkyō City, Tokyo-To
  - Nippon Medical School Hospital, Bunkyō City
  - National Cancer Center Hospital, Chūōku
  - NHO Kyushu Cancer Center, Fukuoka
  - NHO Hokkaido Cancer Center, Hokkaido
  - Cancer Institute Hospital of JFCR, Kōtō City
  - Kurashiki Central Hospital, Kurashiki-shi
  - Kurume University Hospital, Kurume-shi
  - Aichi Cancer Center Hospital, Nagoya
  - NHO Nagoya Medical Center, Nagoya
  - Miyagi Cancer Center, Natori-shi
  - Okayama University Hospital, Okayama
  - Osaka International Cancer Institute, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Osaka
  - Gunma Prefectural Cancer Center, Ota-shi
  - Kanagawa Cancer Center, Yokohama
- Netherlands (9):
  - Amsterdam UMC Locatie VUMC, Amsterdam
  - Antoni van Leeuwenhoek, Amsterdam
  - St. Jansdal Ziekenhuis, Harderwijk
  - Zuyderland Medisch Centrum - Heerlen, Heerlen
  - Leiden University Medical Center, Leiden
  - Radboudumc, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Isala Zwolle, Zwolle
- Poland (5):
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie, Krakow
  - Polish Mother's Memorial Hospital (Instytut Centrum Zdrowia Matki Polki), Lodz
  - Aidport sp z o.o., Skorzewo
  - Instytut Gruzlicy i Chorob Pluc w Warszawie, Warsaw
  - Maria Sklodowska-Curie National Research Institute of Oncology (Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie), Warsaw
- Portugal (4):
  - Unidade Local de Saude de Coimbra E P E, Coimbra
  - Unidade Local de Saúde de Matosinhos, E.P.E. - Hospital Pedro Hispano, Matosinhos Municipality
  - Hospital CUF Porto, Porto
  - Unidade Local de Saude da Arrabida E. P. E, Setúbal
- Puerto Rico (2):
  - Pan American Oncology Trials, LLC, San Juan
  - Auxilio Mutuo Cancer Center, San Juan
- South Korea (7):
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si
  - Keimyung University Dongsan Hospital, Daegu
  - National Cancer Center Korea, Goyang-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (20):
  - ICO l'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba, Córdoba
  - Complejo Hospitalario Universitario de Santiago CHUS, Santiago de Compostela, La Coruña
  - Complejo Hospitalario Universitario Insular Materno-Infantil, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - H.C. Hospitales S.L., Marbella, Málaga
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona
  - ICO Girona, Girona
  - Facility name: Clínica Universidad de Navarra, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Quironsalud Malaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
  - IVO - Instituto Valenciano de Oncologia, Valencia
- Taiwan (5):
  - National Taiwan University Hospital Yunlin Branch, Douliu
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Cancer Center, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital,Linkou, Taoyuan
- Turkey (Türkiye) (9):
  - Adana City Hospital, Adana
  - Medical Park Seyhan Hospital, Adana
  - Ankara City Hospital, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara
  - Gulhane Training and Research Hospital, Ankara
  - Liv Hospital Ankara, Ankara
  - Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - İ.E.Ü. Medicalpoint İzmir Hastanesi, Izmir
- United Kingdom (6):
  - Beatson West of Scotland Cancer Care, Glasgow, Strathclyde
  - Barts Hospital, London
  - Guy's Hospital, London
  - The Christie Hospital, Manchester
  - Nottingham University Hospitals City Campus, Nottingham
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No